CLINICAL TRIAL: NCT07197320
Title: Comparison of Outcomes of Right Internal Jugular Port Implantation in Patients With Right Versus Left Breast Cancer Undergoing Chemotherapy in Gorgan Medical Centers (2017-2024)
Brief Title: Comparison of Outcomes of Right Internal Jugular Port Implantation in Patients With Right Versus Left Breast Cancer Undergoing Chemotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Golestan University of Medical sciences (Other)
Responsible Party: Principal Investigator, Pezhman Kharazm, MD, Assistant Professor of Vascular Surgery, Golestan University of Medical sciences
Other Study IDs: 115103
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Port-A-Cath
Keywords: chemotherapy; port; mastectomy; breast cancer; One-year patency
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients with right-sided breast cancer who received a right internal jugular port
- Cohort 2: Patients with left-sided breast cancer who received a right internal jugular port

SUMMARY:
Chemotherapy is an essential component of breast cancer treatment. Frequent intravenous injections may lead to phlebitis and limited venous access, therefore implantable venous ports are increasingly used. The choice of port placement side in breast cancer patients is controversial, especially when mastectomy or radiotherapy is planned. This retrospective cohort study compares one-year patency, complications (infection, thrombosis, skin necrosis), and functional outcomes of ports implanted via the right internal jugular vein in patients with right versus left breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among women worldwide. Chemotherapy remains a cornerstone of treatment, whether in neoadjuvant or adjuvant settings. Despite advancements in drug formulations, repeated intravenous injections frequently result in phlebitis and loss of venous access. As a result, many patients and physicians prefer the use of totally implantable venous access devices (ports). These devices consist of a catheter and a chamber, allowing direct administration of chemotherapy into a central vein, reducing endothelial damage.

However, ports carry risks including infection, venous thrombosis, skin necrosis, and mechanical failure. In breast cancer patients who undergo mastectomy or radiotherapy, the optimal side for port implantation is controversial. Some surgeons avoid the ipsilateral side due to concerns about complications, while others report no additional risk when proper technique is used.

This retrospective cohort study evaluates the patency and safety of ports implanted through the right internal jugular vein in patients with right- and left-sided breast cancer treated in Gorgan medical centers between 2017 and 2024. Patient records will be reviewed to collect demographic information, tumor laterality, type of breast surgery (mastectomy vs. breast-conserving surgery), use of radiotherapy, type of port, and follow-up outcomes. Complications including infection, thrombosis, and skin necrosis will be recorded. The primary endpoint is one-year port patency; secondary endpoints include complication rates and associations with clinical variables such as age, stage, smoking status, and prior radiotherapy.

This study aims to clarify whether the side of breast cancer affects the outcomes of right internal jugular port implantation, and to provide evidence to guide decision-making regarding optimal port placement in breast cancer patients requiring chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer (right or left side)
* Underwent chemotherapy port implantation via right internal jugular vein between 2017-2024 in Gorgan medical centers

Exclusion Criteria:

* Prior neck surgery or radiotherapy involving right jugular area
* Incomplete medical records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All breast cancer patients receiving right internal jugular venous port implantation in Gorgan medical centers (2017-2024).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
. One-year port patency | 12 months after port implantation
  Defined as functional port access without removal due to complications

SECONDARY OUTCOMES:
Infection | 12 months
  Incidence of port-related infection
Thrombosis | 12 months
  Incidence of port-related thrombosis
skin necrosis | 12 months
  incidence of skin necrosis
cancer side association | 12 months
  Association between port side relative to cancer side and complication rates

CONTACTS AND LOCATIONS:
Locations (1):
- 5Th Azar Medical Center, Gorgan, Outside of the US, Iran

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data will not be shared because of patient privacy concerns and institutional policies.